CLINICAL TRIAL: NCT02413255
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential-Panel, Ascending Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-020 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Single- and Multiple-Doses of TAK-020 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-020-1001; U1111-1163-9637 (Registry Identifier: WHO)
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Part 1 Cohort 1-9: Placebo (Placebo Comparator): TAK-020 placebo-matching solution, orally, once on Day 1.
  Interventions: Drug: TAK-020 Placebo
- Part 1 Cohort 1: TAK-020 0.1 mg (Experimental): TAK-020 0.1 mg, solution, orally once on Day 1.
  Interventions: Drug: TAK-020
- Part 1 Cohort 2: TAK-020 0.5 mg (Experimental): TAK-020 0.5 mg, solution, orally, once on Day 1 following review of safety, tolerability and pharmacokinetic (PK) data from Cohort 1.
  Interventions: Drug: TAK-020
- Part 1 Cohort 3: TAK-020 2.5 mg (Experimental): TAK-020 2.5 mg, solution, orally once on Day 1 following review of safety, tolerability and PK data from Cohort 2.
  Interventions: Drug: TAK-020
- Part 1 Cohort 4: TAK-020 4.4 mg (Experimental): TAK-020 4.4 mg, solution, orally once on Day 1 following review of safety, tolerability and PK data from Cohort 3.
  Interventions: Drug: TAK-020
- Part 1 Cohort 5: TAK-020 8.8 mg (Experimental): TAK-020 8.8 mg, solution, orally once on Day 1 following review of safety, tolerability and PK data from Cohort 4.
  Interventions: Drug: TAK-020
- Part 1 Cohort 6: TAK-020 17.5 mg (Experimental): TAK-020 17.5 mg, solution, orally once on Day 1 following review of safety, tolerability and PK data from Cohort 5.
  Interventions: Drug: TAK-020
- Part 1 Cohort 7: TAK-020 35 mg (Experimental): TAK-020 35 mg, solution, orally once on Day 1. TAK-020 dose will be determined based on review of safety, tolerability and PK data from Cohort 6.
  Interventions: Drug: TAK-020
- Part 1 Cohort 8: TAK-020 70 mg (Experimental): TAK-020 70 mg, solution, orally once on Day 1. TAK-020 dose will be determined based on review of safety, tolerability and PK data from Cohort 7.
  Interventions: Drug: TAK-020
- Part 1 Cohort 9: TAK-020 105 mg (Experimental): TAK-020 105 mg, solution, orally once on Day 1. TAK-020 dose will be determined based on review of safety, tolerability and PK data from Cohort 8.
  Interventions: Drug: TAK-020
- Part 2 Cohort 1-6: Placebo (Placebo Comparator): TAK-020 placebo-matching solution, orally, once on Day 1 and Days 3 to 9.
  Interventions: Drug: TAK-020 Placebo
- Part 2 Cohort 1: TAK-020 3.75 mg (Experimental): TAK-020 3.75 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose are determined based on data from Part 1 of the study.
  Interventions: Drug: TAK-020
- Part 2 Cohort 2: TAK-020 5.75 mg (Experimental): TAK-020 5.75 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose will be determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 1 in Part 2.
  Interventions: Drug: TAK-020
- Part 2 Cohort 3: TAK-020 13 mg (Experimental): TAK-020 13 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose will be determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 2 in Part 2.
  Interventions: Drug: TAK-020
- Part 2 Cohort 4: TAK-020 25 mg (Experimental): TAK-020 25 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose will be determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 3 in Part 2.
  Interventions: Drug: TAK-020
- Part 2 Cohort 5: TAK-020 45 mg (Experimental): TAK-020 45 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose was determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 4 in Part 2.
  Interventions: Drug: TAK-020
- Part 2 Cohort 6: TAK-020 60 mg (Experimental): TAK-020 60 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose was determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 5 in Part 2.
  Interventions: Drug: TAK-020

INTERVENTIONS:
Drug: TAK-020 — TAK-020 oral solution
  Arms: Part 1 Cohort 1: TAK-020 0.1 mg; Part 1 Cohort 2: TAK-020 0.5 mg; Part 1 Cohort 3: TAK-020 2.5 mg; Part 1 Cohort 4: TAK-020 4.4 mg; Part 1 Cohort 5: TAK-020 8.8 mg; Part 1 Cohort 6: TAK-020 17.5 mg; Part 1 Cohort 7: TAK-020 35 mg; Part 1 Cohort 8: TAK-020 70 mg; Part 1 Cohort 9: TAK-020 105 mg; Part 2 Cohort 1: TAK-020 3.75 mg; Part 2 Cohort 2: TAK-020 5.75 mg; Part 2 Cohort 3: TAK-020 13 mg; Part 2 Cohort 4: TAK-020 25 mg; Part 2 Cohort 5: TAK-020 45 mg; Part 2 Cohort 6: TAK-020 60 mg
Drug: TAK-020 Placebo — TAK-020 placebo-matching oral solution
  Arms: Part 1 Cohort 1-9: Placebo; Part 2 Cohort 1-6: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of ascending single- and multiple-doses of TAK-020 in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-020. TAK-020 is being tested to evaluate safety and tolerability of single doses and 7 days multiple doses of TAK-020 in healthy volunteers. This study will look at the PK characteristics (how the drug acts throughout the body) of the drug and safety and tolerability (lab results, vital signs, ECG, and side effects) in healthy participants who take TAK-020.

The study will enroll a total of approximately 120 participants. This study is designed to consist of 2 sequential parts: Part 1-a SRD, and Part 2-a MRD. Healthy participants for Part 1 will be enrolled into 9 cohorts. Each cohort will have 8 randomized participants with receiving a single dose of TAK-020, and 2 receiving matching placebo under fasted conditions. In Cohorts 1-9 doses of 0.1, 0.5, 2.5, 4.4, 8.8, 17.5, 35, 70 and 105 mg will be evaluated.

Healthy participants for Part 2 will be enrolled into 7 cohorts. Each cohort will have 8 randomized participants, with participants receiving one dose of TAK-020 on Day 1, followed by a washout on Day 2, then daily dosing on Days 3-9 of TAK-020 with 2 participants receiving matching placebo under fasted conditions. In Cohorts 1-4 doses of 3.75, 5.75, 13 and 25 mg will be evaluated. For Cohorts 5-7, the subsequent dose level is to be determined based on data from Part 1 and review of safety, tolerability and PK data from Part 2 Cohorts 1-4.

This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 45 days. Participants in Part 1 will make multiple visits to the clinic including a period of confinement to the clinic and will be contacted by telephone 14 days after the last dose of study drug for a follow-up assessment. Participants in Part 2 will make multiple visits to the clinic including a period of confinement to the clinic and will be observed at the clinic 17 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria

Participant eligibility is determined according to the following criteria prior to entry into the study:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. Participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Participant is a healthy adult male or female.
4. The participant is a health adult male or female aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
5. The participant weighs at least 45 kilogram (kg) and has a body mass index (BMI) between 18.0 and 32.0 kilogram per square meter (kg/m^2), inclusive at Screening and Day -1.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use adequate contraception from signing of informed consent throughout the duration of the study and until the next menstrual period or 30 days after last dose, whichever is first. If the next menstrual period is delayed, a pregnancy test will be required for exclusion of pregnancy.

Exclusion Criteria

Any participant who meets any of the following criteria will not qualify for entry into the study:

1. The participant has received any investigational compound within 30 days prior to Screening.
2. The participant is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
3. Participant has a known hypersensitivity to any component of the formulation of TAK-020, Captisol or related compounds.
4. The participant has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
5. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as 4 or more alcoholic beverages per day) within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine.
6. Participant has taken any excluded medication, supplements, or food products, Prohibited Medications and Dietary Products.
7. If female, the participant is pregnant or lactating or intending to become pregnant before, during or within 1 month after exit from this study (30 days post last dose); or intending to donate ova during such time period.
8. If male, the participant intends to donate sperm during the course of this study or for 12 weeks thereafter.
9. Participant has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-020, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
10. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis frequent [more than once per week] occurrence of heartburn, or any surgical intervention [example, cholecystectomy]).
11. Participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
12. Participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day -1).
13. The participant has poor peripheral venous access.
14. Participant has donated or lost 450 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1.
15. Vaccination with any live vaccine within 4 weeks of study drug administration.
16. Participant has a Screening or Check-in (Day -1) abnormal (clinically significant) ECG. Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator medically qualified sub investigator.
17. Participant has QT interval with Fridericia correction method (QTcF) greater than (>) 450 millisecond (msec) for men and women or PR outside the range of 120 to 220 msec confirmed upon repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
18. Participant has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.2* the upper limit of normal (ULN).
    2. Positive screen test for drugs of abuse.
    3. Positive blood screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus-1 or -2 antibodies.
    4. A positive test for tuberculosis (TB) (QuantiFERON).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative sites in the United States from 18 March 2015 to 04 May 2017.
Pre-assignment Details: Healthy volunteers were enrolled to receive TAK-020 oral solution Single Rising Doses (SRD) [0.1, 0.5, 2.5, 4.4, 8.8, 17.5, 35, 70, 105 milligrams (mgs)] or placebo in Part 1 or Multiple Rising Doses (MRD) [3.75, 5.75, 13, 25, 45, 60 mgs] or Placebo in Part 2.
Groups:
- Part 1 Cohort 1: TAK-020 0.1 mg: TAK-020 0.1 milligram (mg), solution, orally once on Day 1.
- Part 1 Cohort 7: TAK-020 35 mg: TAK-020 35 mg, solution, orally once on Day 1. TAK-020 dose was determined based on review of safety, tolerability and PK data from Cohort 6.
- Part 1 Cohort 8: TAK-020 70 mg: TAK-020 70 mg, solution, orally once on Day 1. TAK-020 dose was determined based on review of safety, tolerability and PK data from Cohort 7.
- Part 1 Cohort 9: TAK-020 105 mg: TAK-020 105 mg, solution, orally once on Day 1. TAK-020 dose was determined based on review of safety, tolerability and PK data from Cohort 8.
- Part 2 Cohort 2: TAK-020 5.75 mg: TAK-020 5.75 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose was determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 1 in Part 2.
- Part 2 Cohort 3: TAK-020 13 mg: TAK-020 13 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose was determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 2 in Part 2.
- Part 2 Cohort 4: TAK-020 25 mg: TAK-020 25 mg, solution, orally once on Day 1 and Days 3-9. TAK-020 dose was determined based on data from Part 1 and review of safety, tolerability and PK data from Cohort 3 in Part 2.
Period: Overall Study
Arm/Group | Part 1 Cohort 1-9: Placebo | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg | Part 2 Cohort 1-6: Placebo | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Started | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set was comprised of all participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1-9: Placebo | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg | Part 2 Cohort 1-6: Placebo | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg | Total
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.93) | 46.0 (10.06) | 38.0 (11.15) | 38.0 (11.82) | 29.0 (11.82) | 35.8 (11.44) | 38.2 (12.56) | 33.7 (8.24) | 34.3 (12.61) | 34.8 (7.81) | 37.0 (8.83) | 34.2 (8.59) | 43.2 (9.02) | 29.3 (9.40) | 35.7 (9.40) | 36.2 (11.96) | 34.8 (10.01) | 36.0 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 0 | 3 | 5 | 3 | 3 | 1 | 2 | 0 | 5 | 0 | 3 | 0 | 1 | 1 | 0 | 40
  Male | 7 | 4 | 6 | 3 | 1 | 3 | 3 | 5 | 4 | 6 | 7 | 6 | 3 | 6 | 5 | 5 | 6 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 2 | 2 | 1 | 4 | 3 | 1 | 2 | 0 | 25
  Non-Hispanic and Latino | 16 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 4 | 4 | 10 | 5 | 2 | 3 | 5 | 4 | 6 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 6
  Black or African American | 7 | 4 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 7 | 3 | 1 | 1 | 1 | 1 | 1 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 8 | 2 | 5 | 4 | 5 | 3 | 3 | 4 | 4 | 3 | 5 | 2 | 5 | 4 | 3 | 3 | 4 | 67
  Multiracial | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 120
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 26.18 (3.741) | 27.04 (3.823) | 27.24 (3.308) | 25.77 (4.359) | 23.91 (3.221) | 23.23 (2.549) | 25.87 (3.332) | 23.98 (1.408) | 24.47 (2.263) | 26.89 (1.468) | 25.36 (2.645) | 27.26 (3.516) | 24.97 (4.563) | 25.83 (2.707) | 28.64 (2.935) | 25.07 (2.124) | 27.05 (2.851) | 25.82 (3.223)
Smoking History [Count of Participants; unit: Participants]
  Never Smoked | 16 | 5 | 4 | 6 | 6 | 5 | 4 | 6 | 6 | 5 | 11 | 6 | 4 | 5 | 5 | 6 | 6 | 106
  Ex-smoker | 2 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 14
Alcohol History [Count of Participants; unit: Participants]
  Never drank | 14 | 5 | 6 | 4 | 6 | 6 | 3 | 3 | 4 | 6 | 9 | 4 | 5 | 6 | 4 | 5 | 6 | 96
  Current drinker | 4 | 1 | 0 | 2 | 0 | 0 | 3 | 3 | 2 | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 22
  Ex- drinker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Alcohol Participant Consumed [Count of Participants; unit: Participants] — Number of participants who consume alcohol <4 drinks/day is reported. Population: Assessment was performed on participants who were current drinkers.
  Participants
    number analyzed (Participants) | 4 | 1 | 0 | 2 | 0 | 0 | 3 | 3 | 2 | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 22
    (all) | 4 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 14
Caffeine Consumption [Count of Participants; unit: Participants]
  Yes | 1 | 3 | 1 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 3 | 2 | 2 | 0 | 2 | 2 | 1 | 23
  No | 17 | 3 | 5 | 5 | 5 | 4 | 6 | 6 | 4 | 6 | 9 | 4 | 4 | 6 | 4 | 4 | 5 | 97
Xanthine Consumption [Count of Participants; unit: Participants]
  Yes | 1 | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 3 | 2 | 2 | 0 | 2 | 2 | 1 | 21
  No | 17 | 3 | 5 | 6 | 6 | 4 | 6 | 6 | 4 | 6 | 9 | 4 | 4 | 6 | 4 | 4 | 5 | 99
Female Reproductive Status [Count of Participants; unit: Participants]
  Postmenopausal | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 7
  Surgically Sterile | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4
  Female of Childbearing Potential | 9 | 1 | 0 | 3 | 5 | 2 | 2 | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 29
  Not Applicable (Participant was Male) | 7 | 4 | 6 | 3 | 1 | 3 | 3 | 5 | 4 | 6 | 7 | 6 | 3 | 6 | 5 | 5 | 6 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE) in Part 1 Single-rising Dose (SRD)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event that occurred or worsened after receiving study drug.
Time Frame: First dose of study drug up to and including 30 days after last dose of study drug (Up to 31 days) for Part 1
Population: Safety Analysis Set was comprised of all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1-9: Placebo | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 11.1 | 0 | 0 | 16.7 | 0 | 16.7 | 0 | 0 | 50 | 16.7

2. Primary Outcome: Percentage of Participants With Markedly Abnormal Values (MAV) for Safety Laboratory Findings at Least Once Post-dose in Part 1 (SRD)
Description: Safety laboratory tests includes hematology, serum chemistries, and urinalysis.
Time Frame: From Day 1 to Day 14 of Part 1
Population: Safety Analysis Set was comprised of all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1-9: Placebo | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants
  Hematology | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium <130 mmol/L | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium >150 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin Total >34.2 umol/L | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0
  Triglycerides >2.5*ULN | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (BUN) >10.7 mmol/L | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With MAV for Vital Sign Measurements at Least Once Post-dose in Part 1 (SRD)
Description: Vital signs include oral temperature, respiratory rate, sitting blood pressure (after 5 minutes resting) and pulse beats per minute (bpm).
Time Frame: From Day 1 to Day 14 of Part 1
Population: Safety Analysis Set was comprised of all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1-9: Placebo | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants
  Pulse <50 bpm | 11.1 | 0 | 16.7 | 16.7 | 16.7 | 0 | 0 | 0 | 50 | 0
  Pulse >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure <85 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure >180 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure >110 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Body Temperature <35.6 C | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 16.7
  Body Temperature >37.7 C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With MAV for Safety Electrocardiogram (ECG) Parameters at Least Once Post-dose in Part 1 (SRD)
Description: A standard 12-lead ECG was performed. Change from baseline=CFB.
Time Frame: From Day 1 to Day 14 in Part 1
Population: Safety Analysis Set was comprised of all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1-9: Placebo | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants
  Heart Rate (beats/min) <50 | 44.4 | 16.7 | 16.7 | 50.0 | 16.7 | 16.7 | 0 | 16.7 | 50.0 | 33.3
  Heart Rate (beats/min) >120 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval (msec[ms]) <=80 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval (ms) >= 200 | 5.6 | 0 | 0 | 16.7 | 0 | 16.7 | 16.7 | 50.0 | 0 | 33.3
  QT Interval (ms) <=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval (ms) >=460 | 5.6 | 0 | 16.7 | 33.3 | 16.7 | 16.7 | 0 | 0 | 16.7 | 0
  QTcB Interval (ms) <=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval (ms) ≥500/ ≥30 CFB and ≥450 | 11.1 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 0
  QTcF Interval (ms) <= 300 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval (ms) ≥500/≥30 CFB and >= 450 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Interval (ms) <= 80 | 38.9 | 16.7 | 16.7 | 66.7 | 83.3 | 33.3 | 83.3 | 0 | 16.7 | 50.0
  QRS Interval (ms) >= 180 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE) in Part 2 Multiple-rising Dose (MRD)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event that occurred or worsened after receiving study drug.
Time Frame: First dose of study drug up to and including 30 days after last dose of study drug (Up to 39 days) in Part 2
Population: Safety Analysis Set was comprised of all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1-6: Placebo | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 41.7 | 16.7 | 50.0 | 50.0 | 33.3 | 16.7 | 16.7

6. Primary Outcome: Percentage of Participants With MAV for Safety Laboratory Findings at Least Once Post-dose in Part 2 (MRD)
Description: Safety laboratory tests include hematology, and serum chemistries.
Time Frame: From Day 1 to Day 17 in Part 2
Population: Safety Analysis Set included all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1-6: Placebo | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants
  Hematology | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase >5*ULN (U/L) | 0 | 16.7 | 0 | 0 | 0 | 0 | 16.7
  Lipase >3*ULN (U/L) | 0 | 0 | 0 | 0 | 16.7 | 0 | 0

7. Primary Outcome: Percentage of Participants With MAV for Vital Sign Measurements at Least Once Post-dose in Part 2 (MRD)
Description: Vital signs include oral temperature respiratory rate, sitting blood pressure (after 5 minutes resting) and pulse (bpm).
Time Frame: From Day 1 to Day 17 in Part 2
Population: Safety Analysis Set included all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1-6: Placebo | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants
  Pulse <50 bpm | 8.3 | 0 | 16.7 | 0 | 16.7 | 0 | 16.7
  Pulse >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 16.7
  Systolic Blood Pressure <85 mm Hg | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  Systolic Blood Pressure >180 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 16.7 | 0
  Diastolic Blood Pressure >110 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Body Temperature <35.6 C | 33.3 | 16.7 | 33.3 | 33.3 | 16.7 | 16.7 | 0
  Body Temperature >37.7 C | 0 | 0 | 0 | 0 | 0 | 0 | 16.7

8. Primary Outcome: Percentage of Participants With MAV for Safety ECG Parameters at Least Once Post-dose in Part 2 (MRD)
Description: A standard 12-lead ECG was performed.
Time Frame: From Day 1 to Day 17 in Part 2
Population: Safety Analysis Set included all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1-6: Placebo | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants
  Heart Rate (beats/min) <50 | 16.7 | 16.7 | 16.7 | 50.0 | 50.0 | 16.7 | 16.7
  Heart Rate (beats/min) >120 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval (msec) <=80 | 16.7 | 16.7 | 0 | 0 | 0 | 0 | 0
  PR Interval (msec) >=200 | 16.7 | 16.7 | 0 | 0 | 16.7 | 0 | 16.7
  QT Interval (msec) <=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval (msec) >=460 | 16.7 | 0 | 0 | 16.7 | 33.3 | 16.7 | 16.7
  QTcB Interval (msec) <=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval (ms) ≥500/≥ 30 CFB and ≥450 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval (msec) <=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval (ms) ≥500/≥30 CFB and >= 450 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Interval (msec) <=80 | 50.0 | 33.3 | 50.0 | 16.7 | 0 | 16.7 | 50.0
  QRS Interval (msec) >=180 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-020 in Part 1 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: Pharmacokinetic set included all participants who received study drug and had at least one measurable plasma concentration or amount of drug in the urine.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 0.4631 (36.3) | 1.5529 (25.2) | 13.5475 (40.7) | 24.2013 (29.5) | 42.8329 (43.3) | 105.7708 (33.3) | 155.6549 (31.8) | 446.1922 (50.9) | 345.4612 (51.6)
Statistical Analysis 1: Comparison: Part 1 Cohort 1: TAK-020 0.1 mg vs Part 1 Cohort 2: TAK-020 0.5 mg vs Part 1 Cohort 3: TAK-020 2.5 mg vs Part 1 Cohort 4: TAK-020 4.4 mg vs Part 1 Cohort 5: TAK-020 8.8 mg vs Part 1 Cohort 6: TAK-020 17.5 mg vs Part 1 Cohort 7: TAK-020 35 mg vs Part 1 Cohort 8: TAK-020 70 mg vs Part 1 Cohort 9: TAK-020 105 mg; Test type: Equivalence — Dose proportionality is declared when the 90% confidence interval of the slope lies entirely within the critical region (0.9679, 1.0321) for the dose range of 0.1 mg to 105 mg; p = 0.465, Power Model; Slope = 1.0195, 90% CI 2-sided [0.9752 to 1.0637]

10. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-020 in Part 2 (MRD)
Time Frame: Pre-dose and multiple timepoints (up to 48 hours) post-dose on Day 1 and pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 9 in Part 2
Population: Pharmacokinetic set included all participants who received study drug and had at least one measurable plasma concentration or amount of drug in the urine. Here, number analyzed are the participants who were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  Day 1 | 16.4167 (46.7) | 40.3204 (14.4) | 64.7590 (73.3) | 161.9015 (47.1) | 300.8684 (33.3) | 423.8189 (46.9)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 17.6976 (34.2) | 39.6336 (17.7) | 63.6636 (34.5) | 160.6945 (33.0) | 279.6237 (34.1) | 433.4214 (43.7)
Statistical Analysis 1: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Day 1; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.126, Power Model; Slope = 1.1124, 90% CI 2-sided [0.9913 to 1.2336]
Statistical Analysis 2: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Day 9; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.114, Power Model; Slope = 1.0900, 90% CI 2-sided [0.9962 to 1.1838]

11. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-020 in Part 1 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hr | 0.750 [0.50 to 0.77] | 0.700 [0.48 to 2.02] | 0.745 [0.52 to 1.00] | 0.825 [0.48 to 1.97] | 0.780 [0.67 to 1.05] | 1.010 [0.58 to 2.00] | 0.630 [0.50 to 1.02] | 0.725 [0.50 to 1.00] | 0.750 [0.50 to 2.15]
Statistical Analysis 1: Comparison: Part 1 Cohort 1: TAK-020 0.1 mg vs Part 1 Cohort 2: TAK-020 0.5 mg vs Part 1 Cohort 3: TAK-020 2.5 mg vs Part 1 Cohort 4: TAK-020 4.4 mg vs Part 1 Cohort 5: TAK-020 8.8 mg vs Part 1 Cohort 6: TAK-020 17.5 mg vs Part 1 Cohort 7: TAK-020 35 mg vs Part 1 Cohort 8: TAK-020 70 mg vs Part 1 Cohort 9: TAK-020 105 mg; Test type: Superiority; p = 0.5402, ANOVA; Statistical analysis results were obtained using Analysis of Variance (ANOVA) with dose level as a fixed effect

12. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-020 in Part 2 (MRD)
Time Frame: Pre-dose and multiple timepoints (up to 48 hours) post-dose on Day 1 and pre-dose and multiple time-points (up to 24 hours) post dose on Day 9 in Part 2
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hr
  Day 1 | 0.750 [0.50 to 0.98] | 0.750 [0.52 to 1.08] | 0.750 [0.50 to 2.00] | 0.750 [0.50 to 2.00] | 0.500 [0.50 to 1.02] | 0.640 [0.50 to 1.07]
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 0.750 [0.50 to 1.07] | 1.000 [0.75 to 1.00] | 0.750 [0.50 to 1.00] | 0.750 [0.50 to 0.75] | 0.750 [0.50 to 1.00] | 0.875 [0.47 to 1.98]
Statistical Analysis 1: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Day 1; Test type: Superiority; p = 0.7824, ANOVA; Statistical analysis results were obtained using ANOVA with dose level as a fixed effect
Statistical Analysis 2: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Day 9; Test type: Superiority; p = 0.4056, ANOVA; Statistical analysis results were obtained using ANOVA with dose level as a fixed effect

13. Secondary Outcome: AUC24: Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours for TAK-020 in Part 1 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose in Part 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 0.7599 (45.6) | 3.6691 (28.2) | 29.7502 (48.1) | 63.1772 (31.3) | 98.8228 (34.6) | 272.3381 (39.5) | 372.5881 (35.2) | 1009.0958 (32.3) | 875.0011 (15.9)
Statistical Analysis 1: Comparison: Part 1 Cohort 1: TAK-020 0.1 mg vs Part 1 Cohort 2: TAK-020 0.5 mg vs Part 1 Cohort 3: TAK-020 2.5 mg vs Part 1 Cohort 4: TAK-020 4.4 mg vs Part 1 Cohort 5: TAK-020 8.8 mg vs Part 1 Cohort 6: TAK-020 17.5 mg vs Part 1 Cohort 7: TAK-020 35 mg vs Part 1 Cohort 8: TAK-020 70 mg vs Part 1 Cohort 9: TAK-020 105 mg; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.019, Power Model; Slope = 1.0606, 90% CI 2-sided [1.0187 to 1.1026]

14. Secondary Outcome: AUC24: Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours for TAK-020 in Part 2 (MRD)
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 1 and pre-dose and multiple timepoints (up to 24 hours) post dose on Day 9 in Part 2
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL
  Day 1 | 34.6177 (50.4) | 86.4177 (18.5) | 148.6319 (64.8) | 389.8000 (43.0) | 576.1987 (31.5) | 808.3223 (39.1)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 39.0653 (43.9) | 100.2960 (21.2) | 147.1828 (47.8) | 400.5548 (27.6) | 648.9853 (25.3) | 1011.2702 (44.9)
Statistical Analysis 1: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Day 1; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.258, Power Model; Slope = 1.0789, 90% CI 2-sided [0.9628 to 1.1950]
Statistical Analysis 2: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Day 9; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.144, Power Model; Slope = 1.0929, 90% CI 2-sided [0.9878 to 1.1980]

15. Secondary Outcome: AUC24/D: Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours Divided by TAK-020 Dose for TAK-020 in Part 1 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose in Part 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL/mg | 7.5994 (45.6) | 7.3382 (28.2) | 11.9001 (48.1) | 14.3584 (31.3) | 11.2299 (34.6) | 15.5622 (39.5) | 10.6454 (35.2) | 14.4157 (32.3) | 8.3333 (15.9)

16. Secondary Outcome: AUC24/D: Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours Divided by TAK-020 Dose for TAK-020 in Part 2 (MRD)
Time Frame: Pre-dose and multiple timepoints (up to 24 Hours) post-dose on Day 1 and pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 9 in Part 2
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL/mg
  Day 1 | 9.2314 (50.4) | 15.0292 (18.5) | 11.4332 (64.8) | 15.5920 (43.0) | 12.8044 (31.5) | 13.4720 (39.1)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 10.4174 (43.9) | 17.4428 (21.2) | 11.3218 (47.8) | 16.0222 (27.6) | 14.4219 (25.3) | 16.8545 (44.9)

17. Secondary Outcome: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for TAK-020 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 0.6674 (50.3) | 3.5250 (30.3) | 29.4206 (48.1) | 62.4593 (31.9) | 98.6610 (34.4) | 273.0083 (40.0) | 378.3179 (35.5) | 1024.5599 (32.5) | 903.9858 (14.6)
Statistical Analysis 1: Comparison: Part 1 Cohort 1: TAK-020 0.1 mg vs Part 1 Cohort 2: TAK-020 0.5 mg vs Part 1 Cohort 3: TAK-020 2.5 mg vs Part 1 Cohort 4: TAK-020 4.4 mg vs Part 1 Cohort 5: TAK-020 8.8 mg vs Part 1 Cohort 6: TAK-020 17.5 mg vs Part 1 Cohort 7: TAK-020 35 mg vs Part 1 Cohort 8: TAK-020 70 mg vs Part 1 Cohort 9: TAK-020 105 mg; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.003, Power Model; Slope = 1.0799, 90% CI 2-sided [1.0371 to 1.1227]

18. Secondary Outcome: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for TAK-020 in Part 2 (MRD)
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 34.1425 (50.2) | 85.7708 (18.3) | 148.6319 (64.8) | 391.5478 (43.2) | 583.7178 (32.2) | 823.3525 (39.0)
Statistical Analysis 1: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.201, Power Model; Slope = 1.0897, 90% CI 2-sided [0.9735 to 1.2060]

19. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Calculated Using the Observed Value for the Last Quantifiable Concentration for TAK-020 in Part 1 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 1.3733 (32.1) | 3.8341 (26.8) | 29.9808 (47.4) | 69.3298 (24.2) | 100.2928 (34.3) | 275.1708 (39.6) | 380.2423 (35.2) | 1030.7508 (32.3) | 907.7704 (14.5)
Statistical Analysis 1: Comparison: Part 1 Cohort 1: TAK-020 0.1 mg vs Part 1 Cohort 2: TAK-020 0.5 mg vs Part 1 Cohort 3: TAK-020 2.5 mg vs Part 1 Cohort 4: TAK-020 4.4 mg vs Part 1 Cohort 5: TAK-020 8.8 mg vs Part 1 Cohort 6: TAK-020 17.5 mg vs Part 1 Cohort 7: TAK-020 35 mg vs Part 1 Cohort 8: TAK-020 70 mg vs Part 1 Cohort 9: TAK-020 105 mg; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.490, Power Model; Slope = 1.0188, 90% CI 2-sided [0.9734 to 1.0642]

20. Secondary Outcome: AUC∞:Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Calculated Using the Observed Value for the Last Quantifiable Concentration for TAK-020 in Part 2 (MRD)
Time Frame: Pre-dose and multiple timepoints (up to 48 hours) post-dose on Day 1 in Part 2
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 34.8469 (49.8) | 86.7892 (18.1) | 149.9419 (64.5) | 393.8737 (43.2) | 587.4204 (31.8) | 825.6238 (38.9)
Statistical Analysis 1: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg vs Part 2 Cohort 2: TAK-020 5.75 mg vs Part 2 Cohort 3: TAK-020 13 mg vs Part 2 Cohort 4: TAK-020 25 mg vs Part 2 Cohort 5: TAK-020 45 mg vs Part 2 Cohort 6: TAK-020 60 mg; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.224, Power Model; Slope = 1.0846, 90% CI 2-sided [0.9690 to 1.2002]

21. Secondary Outcome: Rac(AUC): Accumulation Ratio Based on AUC Calculated as AUC24 at Steady State/AUC24 After a Single Dose for TAK-020 (MRD)
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 9 in Part 2
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ratio | 1.1285 (21.9) | 1.1606 (8.9) | 0.9903 (18.7) | 1.0628 (23.3) | 1.1263 (10.7) | 1.2511 (15.6)

22. Secondary Outcome: Rac(Cmax): Accumulation Ratio Based on Cmax Calculated as Cmax at Steady State/Cmax After a Single Dose for TAK-020 (MRD)
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 9 in Part 2
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ratio | 1.0780 (22.9) | 0.9830 (10.5) | 0.9831 (39.4) | 0.9379 (29.2) | 0.9294 (16.3) | 1.0227 (29.5)

23. Secondary Outcome: Cmax/D: Maximum Observed Plasma Concentration Divided by TAK-020 Dose for TAK-020 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL/mg | 4.6312 (36.3) | 3.1058 (25.2) | 5.4190 (40.7) | 5.5003 (29.5) | 4.8674 (43.3) | 6.0440 (33.3) | 4.4473 (31.8) | 6.3742 (50.9) | 3.2901 (51.6)

24. Secondary Outcome: Cmax/D: Maximum Observed Plasma Concentration Divided by TAK-020 Dose for TAK-020 (MRD)
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL/mg
  Day 1 | 4.3778 (46.7) | 7.0123 (14.4) | 4.9815 (73.3) | 6.4761 (47.1) | 6.6860 (33.3) | 7.0636 (46.9)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 4.7194 (34.2) | 6.8928 (17.7) | 4.8972 (34.5) | 6.4278 (33.0) | 6.2139 (34.1) | 7.2237 (43.7)

25. Secondary Outcome: Terminal Disposition Phase Half-life for TAK-020 in Part 1 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hr | 1.1251 (0.16347) | 1.5323 (0.28359) | 2.2093 (0.41162) | 3.0159 (0.70963) | 4.8384 (1.06916) | 4.2946 (1.18227) | 6.0601 (1.55255) | 6.1098 (1.65014) | 9.0275 (4.78526)

26. Secondary Outcome: T1/2z : Terminal Disposition Phase Half-life (T1/2z) for TAK-020 in Part 2 (MRD)
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hr
  Day 1 | 2.5948 (0.42162) | 3.3397 (0.96341) | 4.1895 (0.40518) | 4.8507 (2.21078) | 6.0124 (2.30297) | 6.2971 (1.82711)
  Day 9: number analyzed (Participants) | 4 | 6 | 6 | 5 | 6 | 6
  Day 9 | 2.1537 (0.42833) | 3.2089 (0.77467) | 4.1335 (0.51741) | 3.7934 (0.70657) | 5.1273 (1.58301) | 5.4635 (1.47268)

27. Secondary Outcome: Lambda z (Λz): Terminal Disposition Phase Rate Constant for TAK-020 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
1/hr | 0.6226 (0.09046) | 0.4659 (0.08893) | 0.3223 (0.05573) | 0.2402 (0.05603) | 0.1496 (0.03468) | 0.1745 (0.05957) | 0.1202 (0.02831) | 0.1216 (0.03677) | 0.1004 (0.06068)
Statistical Analysis 1: Comparison: Part 1 Cohort 1: TAK-020 0.1 mg vs Part 1 Cohort 2: TAK-020 0.5 mg vs Part 1 Cohort 3: TAK-020 2.5 mg vs Part 1 Cohort 4: TAK-020 4.4 mg vs Part 1 Cohort 5: TAK-020 8.8 mg vs Part 1 Cohort 6: TAK-020 17.5 mg vs Part 1 Cohort 7: TAK-020 35 mg vs Part 1 Cohort 8: TAK-020 70 mg vs Part 1 Cohort 9: TAK-020 105 mg; Test type: Superiority; p < .0001, ANOVA; Statistical analysis results were obtained using ANOVA with dose level as a fixed effect

28. Secondary Outcome: Lamda z (Λz):Terminal Disposition Phase Rate Constant for TAK-020 (MRD)
Time Frame: From pre-dose to 96 hours post-dose in Part 1 and pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 9 in Part 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
1/hr
  Day 1 | 0.2732 (0.04550) | 0.2231 (0.06562) | 0.1667 (0.01608) | 0.1655 (0.05994) | 0.1263 (0.03599) | 0.1216 (0.04880)
  Day 9: number analyzed (Participants) | 4 | 6 | 6 | 5 | 6 | 6
  Day 9 | 0.3325 (0.07185) | 0.2264 (0.05325) | 0.1699 (0.02117) | 0.1880 (0.03581) | 0.1471 (0.04752) | 0.1363 (0.04310)

29. Secondary Outcome: Tlag: Lag Time to First Quantifiable Concentration for TAK-020 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hr | 0.0000 [0.000 to 0.250] | 0.0000 [0.000 to 0.220] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000]

30. Secondary Outcome: Tlag: Lag Time to First Quantifiable Concentration for TAK-020 (MRD)
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hr
  Day 1 | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000]
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000]

31. Secondary Outcome: CL/F: Apparent Clearance After Extravascular Administration Calculated Using the Observed Value of the Last Quantifiable Concentration of TAK-020 in Part 1 (SRD)
Description: CL/F was calculated as dose/AUC∞.
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h | 74.6058 (22.96089) | 134.3327 (36.96594) | 90.8722 (42.30328) | 64.9449 (15.91608) | 92.1842 (34.02451) | 67.4975 (25.25161) | 96.6058 (32.53095) | 70.7695 (22.35098) | 116.6389 (16.07341)

32. Secondary Outcome: CL/F: Apparent Clearance After Extravascular Administration Calculated Using the Observed Value of the Last Quantifiable Concentration of TAK-020 in Part 2 (MRD)
Description: CL/F was calculated as dose/AUCτ.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
L/h
  Day 1 | 118.3171 (58.62331) | 67.1355 (11.81065) | 100.6915 (62.33954) | 68.2909 (29.74598) | 79.5377 (22.34558) | 76.9650 (28.27771)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 103.2882 (42.85829) | 58.3884 (12.20159) | 96.5521 (46.88638) | 64.1696 (16.00068) | 71.1027 (16.99648) | 64.2873 (29.63651)

33. Secondary Outcome: Apparent Volume of Distribution (Vz/F) During the Terminal Disposition Phase After Extravascular Administration Calculated Using the Observed Value for the Last Quantifiable Concentration for TAK-020 in Part 1 (SRD)
Description: Vz/F was calculated as (CL/F)/λz.
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L | 118.3923 (19.67518) | 292.2714 (78.43782) | 290.5190 (160.50093) | 281.7423 (101.64610) | 655.4794 (320.11459) | 416.8746 (183.79449) | 807.4773 (200.14983) | 594.3399 (149.97225) | 1573.1600 (901.24407)

34. Secondary Outcome: Apparent Volume of Distribution (Vz/F) During the Terminal Disposition Phase After Extravascular Administration Calculated Using the Observed Value for the Last Quantifiable Concentration for TAK-020 in Part 2 (MRD)
Description: Vz/F was calculated as (CL/F)/λz.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
L
  Day 1 | 442.5900 (248.99792) | 329.6057 (135.47030) | 632.4288 (438.98268) | 460.7824 (218.14865) | 698.3679 (373.79793) | 715.0788 (414.96986)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 366.8037 (178.07012) | 266.5672 (68.21454) | 565.3577 (252.08686) | 352.4564 (114.45822) | 530.4696 (211.00235) | 503.3324 (298.76176)

35. Secondary Outcome: Ae(0-24) : Amount of Drug Excreted in Urine During a 24-hour Dosing Interval for TAK-020 in Part 1 (SRD)
Description: Ae(0-24) was calculated as calculated as Cur*Vur, where Cur was the concentration of drug excreted in urine and Vur is the volume of urine excreted.
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg | 0.002473 (0.0008033) | 0.009898 (0.0049671) | 0.069183 (0.0289653) | 0.128195 (0.0412071) | 0.227985 (0.0762743) | 0.507260 (0.1109721) | 0.963253 (0.3108451) | 2.010763 (0.3615714) | 1.925176 (0.6269670)

36. Secondary Outcome: Ae(0-24): Amount of Drug Excreted in Urine During a 24-hour Dosing Interval for TAK-020 in Part 2 (MRD)
Description: Ae(0-24) is calculated as calculated as Cur*Vur, where Cu was the concentration of drug excreted in urine and Vur is the volume of urine excreted.
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 1 and Day 9 in Part 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
mg
  Day 1 | 0.086153 (0.0362135) | 0.149595 (0.0378613) | 0.418761 (0.1666534) | 1.095832 (0.4029873) | 1.186754 (0.3087747) | 1.569498 (0.3542760)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 0.089955 (0.0423540) | 0.181305 (0.0555997) | 0.385163 (0.1034764) | 1.004047 (0.2138181) | 1.370011 (0.3414174) | 2.165337 (0.3525765)

37. Secondary Outcome: Ae(0-96): Amount of Drug Excreted in Urine From Time 0 to Time 96 Hours for TAK-020 in Part 1 (SRD)
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg | 0.002473 (0.0008033) | 0.009999 (0.0049464) | 0.069676 (0.0288376) | 0.128604 (0.0411008) | 0.229946 (0.0763608) | 0.514036 (0.1144776) | 0.977421 (0.3148372) | 2.062580 (0.3829068) | 1.988120 (0.6152605)

38. Secondary Outcome: Fe(0-24): Fraction of Drug Excreted in Urine for TAK-020 in Part 1 (SRD)
Description: Fe was calculated as (Aet/dose)*100.
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of TAK-020 dose
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of TAK-020 dose | 2.4733 (0.80334) | 1.9796 (0.99341) | 2.7673 (1.15861) | 2.9135 (0.93653) | 2.5907 (0.86675) | 2.8986 (0.63413) | 2.7522 (0.88813) | 2.8725 (0.51653) | 1.8335 (0.59711)

39. Secondary Outcome: Fe(0-24): Fraction of Drug Excreted in Urine for TAK-020 in Part 2 (MRD)
Description: Fe was calculated as (Aet/dose)*100.
Time Frame: Pre-dose and multiple timepoints (up to 24 hours) post-dose on Day 1 and Day 9 in Part 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of TAK-020 dose
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
percentage of TAK-020 dose
  Day 1 | 2.2974 (0.96569) | 2.6016 (0.65846) | 3.2212 (1.28195) | 4.3833 (1.61195) | 2.6372 (0.68617) | 2.6158 (0.59046)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 2.3988 (1.12944) | 3.1531 (0.96695) | 2.9628 (0.79597) | 4.0162 (0.85527) | 3.0445 (0.75871) | 3.6089 (0.58763)

40. Secondary Outcome: Fe(0-96): Fraction of Drug Excreted in Urine for TAK-020 in Part 1 (SRD)
Description: Fe was calculated as (Aet/dose)*100.
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of TAK-020 dose
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of TAK-020 dose | 2.4733 (0.80334) | 1.9999 (0.98928) | 2.7870 (1.15351) | 2.9228 (0.93411) | 2.6130 (0.86774) | 2.9373 (0.65416) | 2.7926 (0.89953) | 2.9465 (0.54701) | 1.8934 (0.58596)

41. Secondary Outcome: Renal Clearance (CLr) for TAK-020 in Part 1 (SRD)
Description: CLr was calculated as (Ae96/AUCt)*100.
Time Frame: Pre-dose and multiple timepoints (up to 96 hours) post-dose in Part 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h | 3.6856 (1.20477) | 2.6010 (0.62075) | 2.5250 (1.30987) | 2.0190 (0.47688) | 2.2159 (0.15331) | 1.8896 (0.60426) | 2.6108 (1.03807) | 2.0007 (0.28823) | 2.1898 (0.63728)

42. Secondary Outcome: Renal Clearance (CLr) for TAK-020 in Part 2 (MRD)
Description: CLr was calculated as (Ae24/AUC24)*100.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
L/h
  Day 1 | 2.3165 (0.35669) | 1.7168 (0.42806) | 2.8969 (1.50559) | 2.6497 (0.42235) | 2.1525 (0.83694) | 1.9597 (0.52835)
  Day 9: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
  Day 9 | 2.0802 (0.36760) | 1.7732 (0.41318) | 2.6754 (1.08869) | 2.5311 (0.65737) | 2.2053 (0.80067) | 2.2405 (0.82268)

43. Secondary Outcome: R: Linearity Index Calculated as AUC24 at Steady State/AUC∞ After a Single Dose for TAK-020 in Part 2 (MRD)
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ratio
  Day 1 | 3.551 (0.1578) | 4.463 (0.1578) | 5.010 (0.1578) | 5.940 (0.1728) | 6.376 (0.1578) | 6.716 (0.1578)
  Day 9 | 3.665 (0.1578) | 4.608 (0.1578) | 4.992 (0.1578) | 5.993 (0.1728) | 6.475 (0.1578) | 6.919 (0.1578)
Statistical Analysis 1: Comparison: Part 2 Cohort 1: TAK-020 3.75 mg; Test type: Other; Estimated Ratio = 1.121, 90% CI 2-sided [0.772 to 1.628]
Statistical Analysis 2: Comparison: Part 2 Cohort 2: TAK-020 5.75 mg; Test type: Other; Estimated Ratio = 1.156, 90% CI 2-sided [0.796 to 1.678]
Statistical Analysis 3: Comparison: Part 2 Cohort 3: TAK-020 13 mg; Test type: Other; Estimated Ratio = 0.982, 90% CI 2-sided [0.676 to 1.425]
Statistical Analysis 4: Comparison: Part 2 Cohort 4: TAK-020 25 mg; Test type: Other; Estimated Ratio = 1.055, 90% CI 2-sided [0.701 to 1.587]
Statistical Analysis 5: Comparison: Part 2 Cohort 5: TAK-020 45 mg; Test type: Other; Estimated Ratio = 1.105, 90% CI 2-sided [0.761 to 1.604]
Statistical Analysis 6: Comparison: Part 2 Cohort 6: TAK-020 60 mg; Test type: Other; Estimated Ratio = 1.225, 90% CI 2-sided [0.844 to 1.778]

ADVERSE EVENTS:
Time Frame: First dose of study drug up to and including 30 days after last dose of study drug ( 31 Days for Part 1 and 39 days for Part 2)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 Cohort 1-9: Placebo | Part 1 Cohort 1: TAK-020 0.1 mg | Part 1 Cohort 2: TAK-020 0.5 mg | Part 1 Cohort 3: TAK-020 2.5 mg | Part 1 Cohort 4: TAK-020 4.4 mg | Part 1 Cohort 5: TAK-020 8.8 mg | Part 1 Cohort 6: TAK-020 17.5 mg | Part 1 Cohort 7: TAK-020 35 mg | Part 1 Cohort 8: TAK-020 70 mg | Part 1 Cohort 9: TAK-020 105 mg | Part 2 Cohort 1-6: Placebo | Part 2 Cohort 1: TAK-020 3.75 mg | Part 2 Cohort 2: TAK-020 5.75 mg | Part 2 Cohort 3: TAK-020 13 mg | Part 2 Cohort 4: TAK-020 25 mg | Part 2 Cohort 5: TAK-020 45 mg | Part 2 Cohort 6: TAK-020 60 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/18 | 0/6 | 0/6 | 1/6 | 0/6 | 1/6 | 0/6 | 0/6 | 3/6 | 1/6 | 5/12 | 1/6 | 3/6 | 3/6 | 2/6 | 1/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1-9: Placebo (N=18) | Part 1 Cohort 1: TAK-020 0.1 mg (N=6) | Part 1 Cohort 2: TAK-020 0.5 mg (N=6) | Part 1 Cohort 3: TAK-020 2.5 mg (N=6) | Part 1 Cohort 4: TAK-020 4.4 mg (N=6) | Part 1 Cohort 5: TAK-020 8.8 mg (N=6) | Part 1 Cohort 6: TAK-020 17.5 mg (N=6) | Part 1 Cohort 7: TAK-020 35 mg (N=6) | Part 1 Cohort 8: TAK-020 70 mg (N=6) | Part 1 Cohort 9: TAK-020 105 mg (N=6) | Part 2 Cohort 1-6: Placebo (N=12) | Part 2 Cohort 1: TAK-020 3.75 mg (N=6) | Part 2 Cohort 2: TAK-020 5.75 mg (N=6) | Part 2 Cohort 3: TAK-020 13 mg (N=6) | Part 2 Cohort 4: TAK-020 25 mg (N=6) | Part 2 Cohort 5: TAK-020 45 mg (N=6) | Part 2 Cohort 6: TAK-020 60 mg (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT02413255/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT02413255/SAP_001.pdf